CLINICAL TRIAL: NCT01223898
Title: An Open-label, Two-period, Fixed-sequence Study to Evaluate the Effects of Multiple Doses of Nilotinib on the Pharmacokinetics of Midazolam in CML Patients Who Are Resistant and/or Intolerant Against at Least One Prior Therapy With a BCR-ABL Tyrosine Kinase Inhibitor
Brief Title: To Evaluate the Effects of Multiple Doses of Nilotinib on the Pharmacokinetics and Metabolism of Midazolam in CML Patients With Additional Extension Phase to Evaluate the Safety of Nilotinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAMN107A2128; 2009-009425-28 (EudraCT Number)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML,; nilotinib,; midazolam
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Tasigna

INTERVENTIONS:
Drug: Tasigna
  Other Names: AMN107

SUMMARY:
This study will evaluate the effects of multiple doses of nilotinib on the pharmacokinetics and metabolism of midazolam (as a sensitive CYP3A probe) in CML patients. The following extension study does evaluate the safety of nilotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a cytopathologically confirmed diagnosis of Ph+ CML or Philadelphia chromosome- negative (Ph-) CML patients in accelerated or chronic phase who are resistant and/or intolerant against at least one prior therapy with a BCR-ABL tyrosine kinase inhibitor
2. Female or male ≥ 18 years of age
3. Patients who are nilotinib naïve at study entry, e.g. did not receive any nilotinib treatment prior to study
4. WHO Performance Status of ≤ 2

Exclusion Criteria:

1. Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required).
2. Impaired cardiac function
3. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
4. Patients actively receiving therapy with the prohibited co-medications (CYP3A4 inhibitors or inducers, or CYP2C inducers)
5. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval
6. Treatment with immunotherapy or chemotherapy within 3 days (6 weeks for nitrosurea or mitomycin-C) prior to Day 1 or who have not recovered from side effects of such therapy.
7. Treatment with imatinib within 1 week prior to Day 1 or who have not recovered from side effects of such therapy.
8. Patients who have hypersensitivity to midazolam or related compounds

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
evaluate the effects of multiple doses of nilotinib on the pharmacokinetics and metabolism of midazolam in CML patients. | 2 weeks

SECONDARY OUTCOMES:
evaluate the safety and tolerability of multiple doses of nilotinib when midazolam is co-administered orally in CML patients. | 2 weeks
Monitoring of safety of nilotinib during the extension study phase. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (4):
  - Novartis Investigative Site, Frankfurt/M
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Glasgow, United Kingdom

REFERENCES:
- See also: Results for CAMN107A2128 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12976